CLINICAL TRIAL: NCT04817930
Title: Patient-specific Alloplastic Chin Implant Versus Computer Guided Genioplasty: Soft Tissue Assessment After One Year Follow up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Shawky, Patient-specific Alloplastic Chin Implant Versus Computer Guided Genioplasty: Soft Tissue Assessment After One Year Follow up, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OMFS 3-3-6
Record Dates: First submitted 2021-03-21; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Chin Microgenia
Keywords: Chin microgenia; Orthognathic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient specific chin implant (Experimental): A patient specific chin peek implant was used for chin augmentation
  Interventions: Device: Polyetheretherketone patient specific implant
- computer guided advancement genioplasty (Experimental): Computer guided advancement genioplasty using patient specific cutting and positioning guides
  Interventions: Device: Computer guided advancement genioplasty

INTERVENTIONS:
Device: Polyetheretherketone patient specific implant — a customized peek patient specific implant is place to augment the chin
  Arms: Patient specific chin implant
Device: Computer guided advancement genioplasty — advancement genioplasty using patient specific cutting and positioning surgical stents
  Arms: computer guided advancement genioplasty

SUMMARY:
Two groups with retruded chin skeletal deformity. one treated with patient specific alloplastic implant and the other was treated with computer guided advancement genioplasty. soft tissue assessment was executed after one year

ELIGIBILITY:
Inclusion Criteria:

* Patients whose clinical features revealed possible correction of their facial deformity using chin surgery only
* No prior surgery involving the chin

Exclusion Criteria:

* Patients whose clinical features revealed possible correction of their facial deformity using mandibular surgeries.
* Patients with systemic diseases that carried high risk for general anesthesia.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
soft tissue effect | after one year
  The impact of the interventions on the soft tissue gain after one year

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Shawky, Principal Investigator — Assistant lecturer. OMFS. Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
intervention and effect and demographic data